CLINICAL TRIAL: NCT04923035
Title: Evaluating the Burden of Paediatric Pneumococcal Pneumonia in Malaysia Prior to and During Pneumococcal Conjugate Vaccine (PCV) Implementation
Brief Title: Paediatric Pneumococcal Pneumonia in Malaysia Prior to and During Pneumococcal Conjugate Vaccine (PCV) Implementation
Acronym: MSIP PCV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IMU University, Malaysia (Other)
Collaborators: University of Malaya (Other); Universiti Sains Malaysia (Other); International Islamic University Malaysia (Other); University of Southampton (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Lokman Hakim Sulaiman, MD, Deputy Vice Chancellor Research & Director, Institute of Research, Development and Innovation (IRDI), IMU University, Malaysia
Other Study IDs: MISP #60200
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pneumonia, Pneumococcal; Pneumonia Childhood
Keywords: surveillance; polymerase chain reaction; whole-genome sequencing; pneumococcal urine antigen detection; correlation analysis
MeSH Terms: conditions — Pneumonia, Pneumococcal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab and urine sample for cases and control aged 5 years and below. Nasopharyngeal swab will be cultured and Streptococcus Pneumoniae isolates will be inoculated for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Children aged 5 years and below with clinically diagnosed pneumonia and attending the outpatient's department or admitted as a hospital inpatient at three sentinel sites. Pneumonia. Suspected pneumonia cases will be identified by a family physician or paediatrician based on medical history and clinical symptoms.
  Pneumonia is defined as (WHO Fact Sheet 2019) patient with history of:
  1. cough and/or
  2. difficulty/rapid breathing and/or
  3. intercostal recession,
  4. with or without fever. and supported by chest x-ray findings.
- Control: Healthy children aged 5 years and below without any intercurrent respiratory illness and who is in good health as determined by a brief medical history and/or clinical judgement of the investigator whose parent/LAR is willing and able to give informed consent.

SUMMARY:
The purpose of this research is to provide baseline surveillance of pneumonia in young children in Malaysia before and during the implementation of the pneumococcal conjugate vaccine (PCV). Pneumonia is a respiratory infection that can cause mild to life-threatening disease among all age groups but is the leading infectious cause of death among children globally. The most common cause of pneumonia is infection with a bacteria called Streptococcus pneumoniae, also known as pneumococcus. Hence, immunisation with a pneumococcal vaccine is an effective way to prevent pneumonia. In Malaysia, pneumococcal vaccination under the National Immunisation Programme (NIP) for children has since commenced in December 2020, comprising of 3 doses at four, six and 15 months. The routine use of PCV in children will contribute to reducing the burden of pneumococcal infections in the country, especially severe infections. The ongoing COVID-19 pandemic may also have implications on the pneumococcal serotype and clinical presentation of infections in the community.

DETAILED DESCRIPTION:
This study will be a multi-centre prospective case-control study and the recruitment of clinically diagnosed pneumonia patients and healthy controls aged 5 years and below will be conducted at the three university hospitals; University Malaya Medical Centre (UMMC), Sultan Ahmad Shah Medical Centre@International Islamic University Malaysia (SASMEC@IIUM) and Hospital University Sains Malaysia (HUSM). Subject recruitment and sample collection will be carried out for 24 months. Informed consent and general questionnaire will be administrated by the on-site researchers. Clinical samples will be taken according to approved protocol and local policy to include nasopharyngeal (NP) swab and urine sample. NP swab in a transport medium will be store at -80°C before shipment to the International Medical University (IMU) Advanced Microbiology Collaborative Research Laboratory (AMCRL) in Kuala Lumpur for polymerase chain reaction (PCR) analysis. The data obtained may provide crucial data to support policy decisions on pneumococcal vaccination.

. Specific Objectives

1. To determine the prevalence of Streptococcus pneumoniae (SPN) nasopharyngeal (NP) carriage among children 5 years of age and below with pneumonia and invasive pneumonia disease (IPD) using polymerase chain reaction (PCR) analysis.
2. To determine SPN serotypes in young children during the coronavirus disease 2019 (COVID-19) pandemic by whole-genome sequencing analysis.
3. To identify potential changes in clinical presentation and severity of pneumococcal infection in young children during the COVID-19 pandemic.
4. To evaluate the correlations between SPN serotypes detected in NP carriage and urine sample from the same individual/child.
5. To estimate sensitivity and specificity for SPN serotypes detection in urine among children with pneumonia and IPD.

ELIGIBILITY:
Inclusion Criteria:

- Any child aged 5 years and below who meets the case and control definition and whose parent/legal authorized representative (LAR) is willing to give consent on his/her behalf.

Exclusion Criteria:

* who does not meet the case and control definition
* whose parent/guardian does not give consent on his/her behalf
* who has nasal surgery

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is a prospective case-control study in which all children aged 5 years and below with clinically diagnosed community-acquired pneumonia and healthy controls will be recruited at three study sites. As per assumptions of 95% confidence interval (CI), 80% power and detectable odds ratio (OR) of 1.5, The investigators estimate 164 cases and 164 healthy controls per each sentinel hospital site. Thus, the investigators aim to recruit a total of 500 confirmed pneumonia cases and 500 healthy controls for this study.
Sampling Method: Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Nasopharyngeal (NP) pneumococcal carriages prevalence rate among young children | 24 months
  The absence/presence of nasopharyngeal pneumococcal carriages will be tested using standard bacteriological methods and Streptococcus Pneumoniae (SPN) isolates will be inoculated for DNA extraction and further tested by polymerase chain reaction (PCR) for pneumococcal carriage detection.

SECONDARY OUTCOMES:
Streptococcus pneumoniae (SPN) detection in urine samples among young children | 24 months
  To evaluate the correlations between SPN isolates detected in NP carriage and urine sample from the same individual/child.

CONTACTS AND LOCATIONS:
Overall Officials: Lokman Hakim H Sulaiman, PhD, Principal Investigator — IMU University, Malaysia
Locations (3):
- Malaysia (3):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Sultan Ahmad Shah Medical Centre @International Islamic University Malaysia, Kuantan, Pahang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] La Vincente SF, von Mollendorf C, Ulziibayar M, Satzke C, Dashtseren L, Fox KK, Dunne EM, Nguyen CD, de Campo J, de Campo M, Thomson H, Surenkhand G, Demberelsuren S, Bujinlkham S, Do LAH, Narangerel D, Cherian T, Mungun T, Mulholland EK. Evaluation of a phased pneumococcal conjugate vaccine introduction in Mongolia using enhanced pneumonia surveillance and community carriage surveys: a study protocol for a prospective observational study and lessons learned. BMC Public Health. 2019 Mar 21;19(1):333. doi: 10.1186/s12889-019-6639-y. PMID 30898094
- [Result] Adetifa IMO, Adamu AL, Karani A, Waithaka M, Odeyemi KA, Okoromah CAN, Bello MM, Abubakar IS, Inem V, Scott JAG. Nasopharyngeal Pneumococcal Carriage in Nigeria: a two-site, population-based survey. Sci Rep. 2018 Feb 22;8(1):3509. doi: 10.1038/s41598-018-21837-5. PMID 29472635
- [Derived] Ramzi NH, Hoong ATC, Johari NA, Nathan AM, Teh CSJ, Sulaiman NA, Ilias MI, Deris ZZ, Hazlan SNH, Nasir NSM, Bakar AA, Helmi MAM, Juhari WKW, Kamarudin N, Chong CW, Cleary DW, Clarke SC, Sulaiman LH. Multicentre case-control study of pneumococcal infections among children with pneumonia in Peninsular Malaysia (MY-Pneumo): a study protocol. BMC Public Health. 2024 Aug 20;24(1):2255. doi: 10.1186/s12889-024-19789-9. PMID 39164673